CLINICAL TRIAL: NCT03867877
Title: A Comparison of Daily Undulating Periodization Methods With and Without Functional Exercises in Individuals With Parkinson's Disease
Brief Title: Daily Undulating Periodization Methods With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20181119
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Parkinson Disease; Weight-Lifting Exercise Program
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodized Training with Motor Practice (Experimental): Strength training will use 75-80% of the subject's maximum for the specific exercise and contractions will occur at 2s concentric and 3s eccentric for the strength day. 30-80% of subjects' maximal strength for the power day with high-speed concentric and 2 second eccentric contractions, and exercises that simulate activities of daily living for the motor practice day. All resistance-training will be performed on Keiser air-driven machines. Subjects will perform 10 exercises targeting all major muscle groups. The training will last for 12 consecutive weeks, for a total of 36 visits. Each visit will be approximately 60 minutes long and will consist of 5 minutes warm-up, 50 minutes of training and five minutes of cool-down.
  Interventions: Other: Periodized training with motor practice
- Simple Periodized Training (Experimental): Strength training will use 75-80% of the subject's maximum for the specific exercise and contractions will occur at 2 second concentric and 3 second eccentric for the strength day. 30-80% of subjects' maximal strength for the power day, with high speed concentric and 2 second eccentric contractions, and 60-75% of subjects' maximum strength for the hypertrophy day. All resistance-training will be performed on Keiser air-driven machines. Subjects will perform 10 exercises targeting all major muscle groups. The training will last for 12 consecutive weeks, for a total of 36 visits. Each visit will be approximately 60 minutes long and will consist of 5 minutes warm-up, 50 minutes of training and five minutes of cool-down
  Interventions: Other: Simple Periodized Training

INTERVENTIONS:
Other: Periodized training with motor practice — Exercises at 75-80% of the subject's maximum for strength exercise using contractions with 2 second concentric and 3 second eccentric for the strength day. 30-80% of subjects' maximal strength for the power day with high-speed concentric and 2 second eccentric contractions, and exercises that simulate activities of daily living for the motor practice day. All resistance-training will be performed on Keiser air-driven machines. Subjects will perform 10 exercises targeting all major muscle groups. The training will last for 12 consecutive weeks, for a total of 36 visits. Each visit will be approximately 60 minutes long and will consist of 5 minutes warm-up, 50 minutes of training and five minutes of cool-down.
  Arms: Periodized Training with Motor Practice
Other: Simple Periodized Training — Exercises at 75-80% of the subject's maximum for strength using contractions with 2 second concentric and 3 second eccentric for the strength day. 30-80% of subjects' maximal strength for the power day, with high speed concentric and 2 second eccentric contractions, and for hypertrophy day at 60-75% of subjects' maximum strength. All resistance-training will be performed on Keiser air-driven machines. Subjects will perform 10 exercises targeting all major muscle groups. The training will last for 12 consecutive weeks, for a total of 36 visits. Each visit will be approximately 60 minutes long and will consist of 5 minutes exercise using contractions warm-up, 50 minutes of training and five minutes of cool-down.
  Arms: Simple Periodized Training

SUMMARY:
Compare periodized (cyclic) resistance training with and without motor training specific to activities of daily living.

DETAILED DESCRIPTION:
This study will look at how well two different daily undulating training programs (hypertrophy-strength-power training, versus strength-power-functional training) improve participants' physical functions. All testing procedures will take place at the Max Orovitz Laboratory on the Coral Gables campus. This study will involve a 1-week baseline testing phase, a 2-week familiarization phase, a 9-week intervention phase, and a 1-week post-testing window where subjects must report to the lab for 2 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Hoehn & Yahr Classification of Disability, stage 1-3
* can ambulate with or without an assistive device for at least 50 feet
* able to get up and down from the floor with minimal assistance
* has a score of 24 or above on the Folstein Mini-Mental State Exam

Exclusion Criteria:

* Greater than Stage 3 on the Hoehn & Yahr Classification of Disability
* decline in immune function such as pneumonia or systemic infection
* progressive degenerative disease besides PD
* spinal fusion or other orthopedic surgery in the past six months
* mental disease/psychosis such as dementia
* greater than minimal assistance required for gait and transfers
* inability to make regular time commitments to the scheduled training sessions
* participation in resistance training on a regular basis within the past six months
* inability to provide consent
* pregnancy
* a prisoner

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go Test (TUG) | 2-4 minutes
  The participant will be asked to stand up from a standard chair with a seat height of between 40 and 50 centimeters, walk a 3-meter distance at a normal pace, turn, walk back to the chair, and sit down. The test takes approximately 2-4 minutes to complete with instructions.
Strength Test | 30 minutes
  The participant will perform the concentric phase within the limits of the participant's own specific range of motion for each joint/movement tested over 2 second periods. The tester will gradually increase the resistance for each repetition until the participant are not able to move the lever arm one time through the full range of motion. The participant will be asked how hard the test felt after each repetition and each muscle group will be finished in a maximum of seven repetitions.
Gait Test | 10 minutes
  The gait test will be a standard 10 meter gait test at usual (two trials) and maximum (2 trials) speed. The participant will be timed using a stopwatch.
Seated Medicine Ball Chest Throw | 10 minutes
  Participants will be seated in an armless chair with their backs against the seat back and feet flat on the floor. They will then asked to throw a 3kg medicine ball as far as they can. Subjects are allowed to practice as many times as they want. Two trails will be performed with and a one minute rest will be provided.
30 Second Sit-to-Stand Power Test | 5 minutes
  The participant will be asked to sit in a chair with their feet flat on the ground and their arms placed across their chest. They will stand fully as many times times as they can in 30 seconds.
Mini Best test | 15 minutes
  This is a 14-item test designed to measure the participant's balance while standing still and moving. The test takes about 15-20 minutes and includes the following activities:
  * Sit to stand
  * Rise to toes
  * Stand on one leg
  * Compensatory stepping correction - forward
  * Compensatory stepping correction - backward
  * Compensatory stepping correction - lateral
  * Stance (feet together); eyes open, firm surface
  * Stance (feet together); eyes closed, foam surface
  * Incline eyes closed
  * Change in speed
  * Walk with head turns - horizontal
  * Walk with pivot turns
  * Step over obstacles
  * Timed up and go (TUG) with and without dual task

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Signorile, PhD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Max Orovitz Laboratories, Coral Gables, Florida
  - Max Orovitz Laboratory, Coral Gables, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Strand KL, Cherup NP, Totillo MC, Castillo DC, Gabor NJ, Signorile JF. Periodized Resistance Training With and Without Functional Training Improves Functional Capacity, Balance, and Strength in Parkinson's Disease. J Strength Cond Res. 2021 Jun 1;35(6):1611-1619. doi: 10.1519/JSC.0000000000004025. PMID 33927114